CLINICAL TRIAL: NCT03558503
Title: A Phase 2b, Single-Arm, Multicenter Trial to Evaluate the Efficacy and Safety of UGN-102 as Primary Chemoablative Therapy in Patients With Low Grade (LG) Non-Muscle-Invasive Bladder Cancer (NMIBC) at Intermediate Risk of Recurrence
Brief Title: A Phase 2b Study of UGN-102 for Low Grade Intermediate Risk Non-Muscle-Invasive Bladder Cancer
Acronym: OPTIMA II
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UroGen Pharma Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TC-BC-12
Record Dates: First submitted 2018-05-08; First posted 2018-06-15 (Actual); Results first posted 2022-07-25 (Actual); Last update posted 2022-09-16 (Actual); Status verified 2022-09

CONDITIONS: Bladder Cancer; Urothelial Carcinoma; Urothelial Carcinoma Bladder
Keywords: Non-muscle invasive bladder cancer; Low grade non-muscle invasive bladder cancer; Intermediate risk non-muscle invasive bladder cancer; NMIBC; UGN-102; Mitomycin
MeSH Terms: conditions — Urinary Bladder Neoplasms; Carcinoma, Transitional Cell; Non-Muscle Invasive Bladder Neoplasms | interventions — Mitomycin

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- UGN-102 (Experimental): Patients were treated with 6 once-weekly intravesical instillations of UGN-102.
  Interventions: Drug: UGN-102

INTERVENTIONS:
Drug: UGN-102 — UGN-102 consists of mitomycin and sterile hydrogel (a proprietary thermally responsive gel) that is used to reconstitute mitomycin before instillation. The reverse thermal properties of UGN-102 allow for local administration of mitomycin as a liquid, with subsequent conversion to a semi-solid gel depot following instillation into the bladder.
  The UGN-102 admixture for intravesical instillations contains 75 mg mitomycin in 56 mL admixture (1.33 mg mitomycin per 1 mL).
  Other Names: UGN-102 (mitomycin) for intravesical solution

SUMMARY:
This Phase 2b, single-arm, multicenter study evaluated the efficacy and safety of UGN-102 as primary chemoablative therapy in patients with low grade intermediate risk non-muscle-invasive bladder cancer (LG IR NMIBC).

DETAILED DESCRIPTION:
Eligible patients were treated with 6 once-weekly intravesical instillations of UGN-102.

The ablative effect of UGN-102 was evaluated at the 3-month Visit, which occurred 5 weeks ± 1 week after the last weekly instillation (3 months after initiation of study drug). Response was determined based on visual evaluation by cystoscopy (appearance, number, and size of the lesions) and, if there were remaining lesions, by histopathology of the remaining lesions. Complete response (CR) was defined as having no detectable disease (NDD) and was assessed visually during cystoscopy and also by urine cytology. In the event that the investigator was not sure, and there was suspect tissue, a small biopsy was taken from the suspect tissue to confirm CR in addition to cystoscopy and urine cytology.

Patients who achieved a CR continued to have monthly telephone contacts to document any adverse events (AEs) and changes in concomitant medications and were assessed at 6, 9, and 12 months after the first instillation of UGN-102 for evidence of disease recurrence. Patients who had a non-complete response (non-CR) discontinued the study and continued with standard of care according to their treating physician.

Safety was determined based on a review of AEs, laboratory assessments, and physical examination findings.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to sign an informed consent and comply with the protocol.
2. Has newly diagnosed or historic LG NMIBC (Ta) histologically confirmed by cold cup biopsy at screening or within 6 weeks of screening.
3. Is at intermediate risk of recurrence, defined as having 1 or 2 of the following:

   * Presence of multiple tumors;
   * Solitary tumor > 3 cm;
   * Recurrence (≥ 1 occurrence of LG NMIBC within 1 year of the current diagnosis).
4. Has negative voiding cytology for high grade (HG) disease at or within 6 weeks of enrollment.
5. Willing to use 2 acceptable forms of effective contraception from enrollment through 6 months post treatment if the participant is female or the female partner of a male participant and is of childbearing potential (defined as premenopausal women who have not been sterilized).
6. Has adequate organ and bone marrow function as determined by routine laboratory tests as below:

   * Leukocytes ≥ 3,000 per μL;
   * Absolute neutrophil count ≥ 1,500 per μL;
   * Platelets ≥ 100,000 per μL;
   * Hemoglobin ≥ 9.0 g/dL;
   * Total bilirubin ≤ 1.5 x upper limit of normal (ULN);
   * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 × ULN;
   * Alkaline phosphatase ≤ 2.5 × ULN;
   * Estimated glomerular filtration rate (eGFR) ≥ 30 mL/min.
7. Has no evidence of active urinary tract infection (UTI) at Screening and Baseline visits.

   * In the case of symptomatic UTI, the patient will be treated with a full course of antibiotics, and study drug will be postponed until resolution. In the case of asymptomatic bacteriuria, the use of prophylactic antibiotics and postponement of study drug is left to the discretion of the Principal Investigator (PI).

Exclusion Criteria:

1. History of carcinoma in situ (CIS) on preliminary cystoscopy within 5 years of enrollment.
2. Received Bacillus Calmette-Guérin (BCG) treatment for urothelial carcinoma (UC) within previous 2 years.
3. History of HG papillary UC in the past 2 years.
4. Known allergy or sensitivity to mitomycin.
5. Clinically significant urethral stricture that would preclude passage of a urethral catheter.
6. History of pelvic radiotherapy.
7. History of:

   * Neurogenic bladder;
   * Active urinary retention;
   * Any other condition that would prohibit normal voiding.
8. Past or current muscle invasive (ie, T2, T3, T4) or metastatic UC or concurrent upper tract urothelial carcinoma (UTUC).
9. Has participated in a study with an investigational agent or device within 30 days of enrollment.
10. History of prior treatment with an intravesical chemotherapeutic agent with the exception of a single dose of chemotherapy immediately after any previous transurethral resection of bladder tumors (TURBT).
11. Has an underlying substance abuse or psychiatric disorder such that, in the opinion of the investigator, the patient would be unable to comply with the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2018-10-15 (Actual); Primary Completion 2020-01-03 (Actual); Study Completion 2020-10-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elyse Seltzer, MD, Study Director — UroGen Pharma
Locations (19):
- United States (17):
  - Mayo Clinic Cancer Center, Phoenix, Arizona
  - Arkansas Urology, Little Rock, Arkansas
  - Loma Linda University, Loma Linda, California
  - Providence Medical Institute, Santa Monica, California
  - Clinical Research Center of Florida, Pompano Beach, Florida
  - John Hopkins University, Baltimore, Maryland
  - Adult & Pediatric Urology, PC, Omaha, Nebraska
  - Urology Las Vegas, Las Vegas, Nevada
  - Manhattan Medical Research, New York, New York
  - Weill Cornell Medical College, New York, New York
  - Montefiore Medical Center (Albert Einstein), New York, New York
  - Western New York Urology Associates, New York, New York
  - The University of North Carolina, Chapel Hill, North Carolina
  - Penn State Hershey State College, Hershey, Pennsylvania
  - Carolina Urologic Research Center, Myrtle Beach, South Carolina
  - Urology Associates, PC, Nashville, Tennessee
  - Urology San Antonio, Fredericksburg, Texas
- Israel (2):
  - Carmel Medical Center, Haifa
  - Rabin Medical Center, Petah Tikva

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Chevli KK, Shore ND, Trainer A, Smith AB, Saltzstein D, Ehrlich Y, Raman JD, Friedman B, D'Anna R, Morris D, Hu B, Tyson M, Sankin A, Kates M, Linehan J, Scherr D, Kester S, Verni M, Chamie K, Karsh L, Cinman A, Meads A, Lahiri S, Malinowski M, Gabai N, Raju S, Schoenberg M, Seltzer E, Huang WC. Primary Chemoablation of Low-Grade Intermediate-Risk Nonmuscle-Invasive Bladder Cancer Using UGN-102, a Mitomycin-Containing Reverse Thermal Gel (Optima II): A Phase 2b, Open-Label, Single-Arm Trial. J Urol. 2022 Jan;207(1):61-69. doi: 10.1097/JU.0000000000002186. Epub 2021 Aug 26. PMID 34433303
- [Derived] Prasad SM, Louie MJ, Burger B, Tsurutis V, Ugwuoke N, Strauss-Ayali D. Pharmacokinetics of UGN-102, an investigational mitomycin-containing reverse thermal gel for the treatment of non-muscle invasive bladder cancer. Cancer Chemother Pharmacol. 2025 Oct 11;95(1):100. doi: 10.1007/s00280-025-04821-5. PMID 41074972
- [Derived] Stover AM, Basak R, Mueller D, Lipman R, Teal R, Hilton A, Giannone K, Waheed M, Smith AB. Minimal Patient-Reported Side Effects for a Chemoablative Gel (UGN-102) Used as Frontline Treatment in Adults with Nonmuscle-Invasive Bladder Cancer. J Urol. 2022 Sep;208(3):580-588. doi: 10.1097/JU.0000000000002747. Epub 2022 May 31. PMID 35640276

RESULTS

PARTICIPANT FLOW:
Groups:
- UGN-102: 6 once-weekly intravesical instillations of UGN-102.
Period: Overall Study
Arm/Group | UGN-102
Started | 63
Completed | 60
Not Completed | 3
Not completed — Adverse Event | 1
Not completed — Death | 1
Not completed — Refused to come in for the final 12-month assessment due to COVID-19 | 1

BASELINE CHARACTERISTICS:
Arm/Group | UGN-102
Number analyzed (Participants) | 63
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 27
  >=65 years | 36
Age, Continuous [Median (Full Range); unit: years] | 68 [33 to 96]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25
  Male | 38
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 55
  African American | 1
  Hispanic | 3
  Asian | 3
  Other | 1
Tumor Size [Count of Participants; unit: Participants] — Population: Data on tumor size were missing for 2 patients.
  Participants
    number analyzed (Participants) | 61
    <=3 centimeters | 44
    >3 centimeters | 17
Tumor Number [Count of Participants; unit: Participants] — Population: Data on tumor number were missing for 2 patients.
  Participants
    number analyzed (Participants) | 61
    Single | 11
    Multiple | 50
Visual Appearance of Lesions [Number; unit: participants] — Patients may be included in more than one category of visual appearance of lesions.
  participants
    Papillary | 63
    Flat | 2
    Other | 2
Tumor Staging [Number; unit: participants] — Patients may be included in more than one category of tumor staging.
  participants
    Noninvasive papillary carcinoma | 62
    Other | 2
Tumor Grading [Number; unit: participants] — Patients may be included in more than one category of tumor grading.
  participants
    Papillary urothelial carcinoma, low grade | 62
    Papillary urothelial neoplasm of low malignant potential | 1
    Other | 2
Any Previous Low Grade Non-muscle-invasive Bladder Cancer (LG NMIBC) Episode [Count of Participants; unit: Participants]
  Yes | 49
  No | 14
Previous LG NMIBC Episode Within 1 Year of Current Diagnosis [Count of Participants; unit: Participants]
  Yes | 28
  No | 35
Number of Previous LG NMIBC Episodes [Count of Participants; unit: Participants]
  0 | 14
  1-2 | 17
  >2 | 32
Number of Prior Transurethral Resection of Bladder Tumors (TURBT) [Mean (Full Range); unit: TURBTs] — Population: Data on prior TURBT were summarized for patients with a previous LG NMIBC episode.
  TURBTs
    number analyzed (Participants) | 49
    (all) | 4 [0 to 13]
Patients With Number of Prior TURBT [Count of Participants; unit: Participants] — Population: Data on prior TURBT were summarized for patients with a previous LG NMIBC episode.
  Participants
    number analyzed (Participants) | 49
    0 | 2
    1 | 10
    2 | 9
    >=3 | 28
Days Since Last TURBT at Time of Day 1 [Count of Participants; unit: Participants] — Population: Days since last TURBT were summarized for patients with a previous LG NMIBC episode and a prior TURBT.
  Participants
    number analyzed (Participants) | 47
    <=365 | 23
    >365 | 24

OUTCOME MEASURES:

1. Primary Outcome: Complete Response (CR) Rate for UGN-102 Treatment
Description: To evaluate the tumor ablative effect of UGN-102 in patients with LG NMIBC. CR rate was defined as the percentage of patients with no detectable disease (NDD) as determined by cystoscopy, for cause biopsy, and urine cytology.
Time Frame: 3 months after the first instillation of UGN-102
Population: Intent-to-treat (ITT) analysis set (all patients who were enrolled into the study and received at least one instillation of UGN-102)
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | UGN-102
Number analyzed (Participants) | 63
percentage of patients | 65.1 [52.0 to 76.7]

2. Secondary Outcome: Durable Complete Response (DCR) Rate
Description: To evaluate the durability of response in patients with LG NMIBC who achieve CR. DCR rate was defined as the percentage of patients who maintained CR at the respective time point.
Time Frame: 6, 9, and 12 months after the first instillation of UGN-102
Population: 3-month CR analysis set (patients who achieved CR at the 3-month Visit)
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | UGN-102
Number analyzed (Participants) | 41
percentage of patients
  6 months (3 months after CR at the 3-month Visit) | 95.1 [83.5 to 99.4]
  9 months (6 months after CR at the 3-month Visit) | 73.2 [57.1 to 85.8]
  12 months (9 months after CR at the 3-month Visit) | 61.0 [44.5 to 75.8]

3. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs), Study Drug or Procedure Related TEAEs, TEAEs by Maximum Severity, TEAEs Leading to Treatment Discontinuation, and Serious TEAEs.
Description: The number of patients with each type of event will be summarized. Adverse event severity was graded according to Common Terminology Criteria for Adverse Events version 5.0 as follows: Grade 1 (mild), Grade 2 (moderate), Grade 3 (severe or medically significant), Grade 4 (life-threatening), Grade 5 (fatal).
Time Frame: Up to 12 months
Population: ITT analysis set (all patients who were enrolled into the study and received at least one instillation of UGN-102), which is identical to the safety analysis set for this study
Measure: Count of Participants; unit: Participants
Arm/Group | UGN-102
Number analyzed (Participants) | 63
Participants
  Any TEAEs | 57
  Any study drug or procedure related TEAEs | 40
  Maximum severity Grade 1 | 26
  Maximum severity Grade 2 | 24
  Maximum severity Grade 3 | 5
  Maximum severity Grade 4 | 1
  Maximum severity Grade 5 | 1
  Any TEAEs leading to treatment discontinuation | 6
  Any serious TEAEs | 5

4. Secondary Outcome: Number of Participants With Post-baseline Potentially Clinically Significant (PCS) Laboratory Values
Description: The number of patients who met PCS criteria for chemistry or hematology parameters post-baseline will be summarized
Time Frame: Up to 12 months
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | UGN-102
Number analyzed (Participants) | 63
Participants
  Any PCS chemistry value | 8
  Any PCS hematology value | 4

5. Secondary Outcome: Number of Participants With Post-baseline PCS Vital Signs Values
Description: The number of patients who met PCS criteria for vital signs parameters post-baseline will be summarized
Time Frame: Up to 12 months
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | UGN-102
Number analyzed (Participants) | 63
Participants | 8

6. Secondary Outcome: Number of Participants With Post-baseline Clinically Significant (CS) Physical Examination Findings
Description: The number of patients with abnormal, CS physical examination findings post-baseline will be summarized
Time Frame: Up to 12 months
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | UGN-102
Number analyzed (Participants) | 63
Participants | 0

7. Secondary Outcome: Number of Participants With Post-baseline CS Urology-oriented Physical Examination Findings
Description: The number of patients with abnormal, CS urology-oriented physical examination findings post-baseline will be summarized
Time Frame: Up to 12 months
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | UGN-102
Number analyzed (Participants) | 63
Participants | 2

8. Other Pre Specified Outcome: Mitomycin Plasma Concentrations
Description: Mitomycin plasma concentrations were assessed in a subset of 6 patients treated with UGN-102
Time Frame: 0 (pre-instillation), 0.5, 1, 2, 3, 4, 5, and 6 hours after the first instillation of UGN-102
Population: Pharmacokinetic (PK) analysis set (all patients who consented to provide blood samples for PK analysis and had at least 1 plasma sample for evaluation of PK properties of mitomycin following an initial instillation of UGN-102)
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | UGN-102
Number analyzed (Participants) | 6
ng/mL
  Pre-instillation | 0 (0)
  0.5 hours post-instillation | 0.75 (0.57)
  1 hour post-instillation | 0.60 (0.42)
  2 hours post-instillation | 0.34 (0.17)
  3 hours post-instillation | 1.88 (3.13)
  4 hours post-instillation | 1.93 (3.49)
  5 hours post-instillation | 0.57 (0.61)
  6 hours post-instillation | 0.32 (0.32)

9. Other Pre Specified Outcome: Mitomycin Area Under the Plasma Concentration-time Curve (AUC)
Description: Mitomycin AUC was assessed in a subset of 6 patients treated with UGN-102
Time Frame: 0 (pre-instillation) to 6 hours after the first instillation of UGN-102
Population: PK analysis set (all patients who consented to provide blood samples for PK analysis and had at least 1 plasma sample for evaluation of PK properties of mitomycin following an initial instillation of UGN-102)
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | UGN-102
Number analyzed (Participants) | 6
ng*h/mL | 5.69 (7.30)

10. Other Pre Specified Outcome: Mitomycin Maximum Plasma Concentration (Cmax)
Description: Mitomycin Cmax was assessed in a subset of 6 patients treated with UGN-102
Time Frame: 0 (pre-instillation), 0.5, 1, 2, 3, 4, 5, and 6 hours after the first instillation of UGN-102
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | UGN-102
Number analyzed (Participants) | 6
ng/mL | 2.27 (3.33)

ADVERSE EVENTS:
Time Frame: Up to 12 months
Arm/Group | UGN-102
All-Cause Mortality (participants affected / at risk) | 1/63
Serious Adverse Events (participants affected / at risk) | 5/63
Other Adverse Events (participants affected / at risk) | 57/63
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | UGN-102 (N=63)
Acute myeloid leukemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Gastroenteropancreatic neuroendocrine tumor disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Transitional cell carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cardiac disorder (Cardiac disorders) | 1
Stress cardiomyopathy (Cardiac disorders) | 1
Pneumonia (Infections and infestations) | 1
Pneumonia klebsiella (Infections and infestations) | 1
Hematuria (Renal and urinary disorders) | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | UGN-102 (N=63)
Dysuria (Renal and urinary disorders) | 26
Pollakiuria (Renal and urinary disorders) | 13
Hematuria (Renal and urinary disorders) | 9
Micturition urgency (Renal and urinary disorders) | 9
Urinary tract infection (Renal and urinary disorders) | 9
Urinary incontinence (Renal and urinary disorders) | 5
Nocturia (Renal and urinary disorders) | 4
Urinary retention (Renal and urinary disorders) | 4
Pruritus genital (Reproductive system and breast disorders) | 4
Vulvovaginal discomfort (Reproductive system and breast disorders) | 4
Fatigue (General disorders) | 7
Accidental exposure to product (Injury, poisoning and procedural complications) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-04-15): https://cdn.clinicaltrials.gov/large-docs/03/NCT03558503/Prot_000.pdf
  • Statistical Analysis Plan (2020-07-24): https://cdn.clinicaltrials.gov/large-docs/03/NCT03558503/SAP_001.pdf